CLINICAL TRIAL: NCT00210379
Title: A Phase II Study of CHOP + Rituximab, With Intrathecal Methotrexate Followed by Radiotherapy in Patients With Primary Testicular Non-Hodgkin's Lymphoma
Brief Title: Phase II Study of Combined Modality Treatment in Primary Testicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: International Extranodal Lymphoma Study Group (IELSG), IELSG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG10
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Lymphoma, B Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab; Radiotherapy

INTERVENTIONS:
Drug: rituximab
Drug: CHOP
Drug: intrathecal methotrexate
Procedure: radiotherapy

SUMMARY:
The primary objective assess the clinical activity of combination doxorubicin-containing chemotherapy plus monoclonal antibody anti-CD20 (Rituximab) plus intrathecal prophylactic chemotherapy and loco-regional radiotherapy in primary localised testicular DLCL and to assess the toxicity of this therapeutic strategy

ELIGIBILITY:
Inclusion Criteria:

1. age = 18 years.
2. ECOG performance status 0-2
3. Histologically proven primary testicular CD20-positive diffuse large B-cell non-Hodgkin's lymphoma, untreated
4. Ann Arbor stage IE or IIE. Bilateral testicular involvement at presentation will not be considered stage IV. In these patients the final Ann Arbor stage will be determined by the extent of nodal involvement.
5. Bidimensionally measurable or evaluable disease. Patients who have had all disease removed by surgery are eligible.
6. Adequate bone marrow reserve (ANC > 1.000/L, Plt > 100.000/L)
7. Cardiac ejection fraction ≥ 50% by MUGA scan or echocardiography
8. No previous therapy with monoclonal antibody anti-CD20.
9. No psychiatric illness that precludes understanding concepts of the trial or signing informed consent
10. No other major life-threatening illnesses that may preclude chemotherapy
11. Have given written informed consent prior to any program-specific screening procedure, with the understanding that the consent may be withdrawn by the patient at any time without prejudice

Exclusion Criteria:

1. impairment of renal function (creatinine > 2 mg/dl) or liver function (bilirubin > 2 mg/dl) unless due to lymphoma involvement
2. HIV positive patients
3. evolutive malignancy within 5 years with the exception of localized non-melanomatous skin cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2000-11; Primary Completion 2004-11 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Disease-free survival
Progression-free survival
Event-free survival

SECONDARY OUTCOMES:
Overall survival will be a secondary end-point because post-relapse therapy is not specified in this protocol and is expected to be highly variable

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Sarris, MD, Study Chair — International Extranodal Lymphoma Study Group; Emanuele Zucca, MD, Study Chair — International Extranodal Lymphoma Study Group/Oncology Institute of Southern Switzerland (IOSI); Mary Gospodarowicz, MD, Study Chair — Radiation Oncology. Princess Margareth Hospital. Toronto; Umberto Vitolo, MD, Study Chair — Hematology Division. Ospedale San Giovanni Battista. Torino
Locations (1):
- Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Switzerland

REFERENCES:
- See also: Click here for more information about this study — http://www.ielsg.org